CLINICAL TRIAL: NCT01602237
Title: Preventing Respiratory Health Problems in Bakery Employees.
Acronym: Baker2012
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/2449
Record Dates: First submitted 2012-03-05; First posted 2012-05-18 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Lung Disease; Rhinitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Rhinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum, Nasal lavage fluid (without cells)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bakery workers

SUMMARY:
The study is a follow-up of investigations done in the years 1999-2002 in bakery employees. The main purposes are to look at the associations between flour dust exposure and respiratory disease, and to find out the best ways to reduce the flour dust levels in the working environment.

DETAILED DESCRIPTION:
Background and Methods:

Supported by the The Confederation of Norwegian Enterprise (CNBI) Working Environment Fund a follow-up study of 184 bakery workers in 5 bakeries was done in 2012, appr. 10 years after a similar study in 1999-2002. In addition a cross-sectional study in 2 other bakeries (one 'bread-factory', and a traditional bakery with three small bake shops) was added.

Altogether 253 participants, among them 61 former bakery workers, were investigated with use of questionnaires, allergy-testing (skin prick testing, and blood samples for specific IgE and total IgE), spirometry with reversibility testing, exhaled NO-measurement, and nasal measurements.

As in 1999-2002 an extensive exposure assessment was performed including personal samples of total dust (Gelman), inhalable dust (PAS6), as well as direct reading measurements of dust (Dust Track). A Job Exposure Matrix (JEM) was created enabling each participant to be assigned an exposure value of probable mean daily flour-dust exposure based on work-tasks and bakery.

Aim of study:

* Follow-up of the participants in the 1999-2002 study, both still active bakery workers and former workers, on health-status focusing on respiratory disease, sensitization to common and occupational allergens, level of sick-leave and reasons for quitting as a baker.
* Inclusion of 'new' bakery workers into the cohort as a cross-sectional study, and to compare health-status in two cross-sectional cohorts.
* To assess personal exposure to flour-dust among workers in 7 bakeries, as part of the cross-sectional study described above.
* To identify implemented flour-dust exposure reduction measures in bakeries participating in 1999-2002, and to assess the potential impact of these measures on the exposure to flour dust.

ELIGIBILITY:
Inclusion Criteria:

* Employed in a bakery for more than 6 months
* and/or participant of the investigations done in 1999-2002 in 6 bakeries

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. All the employees in 5 bakeries investigated in 1999-2002 (one of the original 6 bakeries has fused with one of the others)
  2. All the employees in additional 2 bakeries located in the same Hordaland county, Norway, as the other 5 bakeries
Sampling Method: Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Forced Exhaled Volume in one second (FEV1) | Change/decline from 1999-2002 to 2012
  The decline in FEV1 from 1999-2002 to 2012.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | Each participant will be investigated once. Anticipated recruitment time for the whole cohort (study population I and II): about 10 months.
  Before and after salbutamol-inhalation. Post-bronchodilatory measurements of FEV1 and FVC to measure the prevalence of chronic obstructive lung disease in a cohort of bakery workers
Inflammation markers in nasal lavage | Each participant will be investigated once. Anticipated recruitment time for the whole cohort (study population I and II): about 10 months.
  Measurement in nasal lavage of inflammation markers (albumin, tryptase, eosinophilic cationic protein) when at work (field study)
Specific IgE | Each participant will be investigated once. Anticipated recruitment time for the whole cohort (study population I and II): about 10 months.
  In serum measurement of specific IgE to common airborne allergens, and allergens mainly found in bakeries
Skin reaction to prick testing with allergen extracts | Each participant will be investigated once. Anticipated recruitment time for the whole cohort (study population I and II): about 10 months.
  Skin prick test with commercially available allergen extracts (common and occupational allergens in bakeries)

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir Storaas, PhD, MD, Principal Investigator — Haukeland University Hospital; Tor B Aasen, MD, Study Director — Haukeland University Hospital
Locations (1):
- Dept. of Occupational Medicine, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Background] Storaas T, Irgens A, Florvaag E, Steinsvag SK, Ardal L, Do TV, Greiff L, Aasen TB. Bronchial responsiveness in bakery workers: relation to airway symptoms, IgE sensitization, nasal indices of inflammation, flour dust exposure and smoking. Clin Physiol Funct Imaging. 2007 Sep;27(5):327-34. doi: 10.1111/j.1475-097X.2007.00755.x. PMID 17697030
- [Background] Storaas T, Ardal L, Van Do T, Florvaag E, Steinsvag SK, Irgens A, Aasen TB, Greiff L. Nasal indices of eosinophilic and exudative inflammation in bakery-workers. Clin Physiol Funct Imaging. 2007 Jan;27(1):23-9. doi: 10.1111/j.1475-097X.2007.00707.x. PMID 17204034
- [Background] Storaas T, Steinsvag SK, Florvaag E, Irgens A, Aasen TB. Occupational rhinitis: diagnostic criteria, relation to lower airway symptoms and IgE sensitization in bakery workers. Acta Otolaryngol. 2005 Nov;125(11):1211-7. doi: 10.1080/00016480510044205. PMID 16353405
- [Result] Kirkeleit J, Hollund BE, Riise T, Eduard W, Bratveit M, Storaas T. Bakers' exposure to flour dust. J Occup Environ Hyg. 2017 Feb;14(2):81-91. doi: 10.1080/15459624.2016.1225156. PMID 27540715